CLINICAL TRIAL: NCT00483470
Title: Immunogenicity and Safety of Sanofi Pasteur's AVAXIM 80U Pediatric Vaccine Followed by Booster Dose
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HAF78
Record Dates: First submitted 2007-06-05; First posted 2007-06-07 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Hepatitis A
Keywords: Hepatitis A
MeSH Terms: conditions — Hepatitis A | interventions — Hepatitis A Vaccines

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: Hepatitis A vaccine AVAXIM 80U
- 2 (Active Comparator)
  Interventions: Biological: Hepatitis A vaccine (HAVRIX 720)

INTERVENTIONS:
Biological: Hepatitis A vaccine AVAXIM 80U — 0.5 mL, Intramuscular
  Other Names: AVAXIM 80U Pediatric vaccine
  Arms: 1
Biological: Hepatitis A vaccine (HAVRIX 720) — 0.5 mL, Intramuscular
  Arms: 2

SUMMARY:
As per request by the Heath Authorities, the present clinical study will assess the immunogenicity and safety

ELIGIBILITY:
Inclusion Criteria :

Inclusion criteria to be checked at the screening visit (SC):

1. Toddlers, children and adolescents:

   Sub-Group 1: from 12 months to 3 years of age on the day of inclusion

   Sub-Group 2: from 4 to 6 years of age on the day of inclusion

   Sub-Group 3: from 7 to 9 years of age on the day of inclusion

   Sub-Group 4: from 10 to 12 years of age on the day of inclusion

   Sub-Group 5: from 13 to 15 years of age on the day of inclusion
2. Screening informed consent form signed by the parent(s) or other legal representative for all the subjects and by the adolescents (sub-group 5 only)

Inclusion criteria to be checked at the inclusion visit (V01):

1. Toddlers, children and adolescents:

   Sub-Group 1: from 12 months to 3 years of age on the day of inclusion

   Sub-Group 2: from 4 to 6 years of age on the day of inclusion

   Sub-Group 3: from 7 to 9 years of age on the day of inclusion

   Sub-Group 4: from 10 to 12 years of age on the day of inclusion

   Sub-Group 5: from 13 to 15 years of age on the day of inclusion
2. Inclusion informed consent form signed by the parent(s) or other legal representative for all the subjects and by the adolescents (sub-group 5 only)
3. Able to attend all scheduled visits and to comply with all trial procedures
4. Subject anti-HAV seronegative (IgG) according to the screening results (assay performed with local kit)
5. Subject HBsAg seronegative and ALT <40 IU/l according to the screening results

Exclusion Criteria :

Exclusion criteria to be checked at the inclusion visit (V01):

1. Participation in another clinical trial in the 4 weeks preceding trial vaccination
2. Planned participation in another clinical trial during the present trial period
3. Congenital or acquired immunodeficiency, immunosuppressive therapy such as long-term systemic corticosteroids therapy
4. Systemic hypersensitivity to any of the vaccines components or history of a life-threatening reaction to the trial vaccines or a vaccine containing the same substances
5. Chronic illness at a stage that could interfere with trial conduct or completion
6. Blood or blood-derived products received in the past 3 months
7. Any vaccination in the 4 weeks preceding the trial vaccination
8. Any vaccination planned in the 4 weeks following the trial vaccination
9. History of hepatitis A infection (confirmed either clinically or serologically )
10. Previous vaccination against hepatitis A with the trial vaccine or another hepatitis A vaccine
11. Thrombocytopenia or a bleeding disorder contraindicating intramuscular vaccination
12. History of /current seizures
13. Clinical or serological evidence of systemic illness including Hepatitis C and HIV
14. Febrile (axillary temperature ≥ 37.1°C) or acute illness

Ages: 12 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 720 (Actual)
Dates: Start 2007-06; Primary Completion 2008-05 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the immunogenicity of AVAXIM 80U Pediatric vaccine | 1 month post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc
Locations (3):
- China (3):
  - Guilin, Guangxi
  - Nanning, Guangxi
  - Yongfu Country, Guangxi

REFERENCES:
- [Derived] Yoon SH, Kim HW, Ahn JG, Kim IT, Kim JH, Kong KA, Kim KH. Reappraisal of the Immunogenicity and Safety of Three Hepatitis A Vaccines in Adolescents. J Korean Med Sci. 2016 Jan;31(1):73-9. doi: 10.3346/jkms.2016.31.1.73. Epub 2015 Dec 24. PMID 26770041
- See also: Related Info — http://www.sanofipasteur.com